CLINICAL TRIAL: NCT04898751
Title: Analysis of Reporting of Cutaneous Toxicities Associated With Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: JH IRB00210048
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Cutaneous Toxicity From ICI Therapy
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Ipilimumab; Nivolumab; pembrolizumab; durvalumab; avelumab; atezolizumab; cemiplimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cutaneous toxicity: Patients who reported a cutaneous immune related adverse event following ICI initiation with appropriate chronology that indicates drug toxicity.
  Interventions: Drug: Immune checkpoint inhibitor (ICI)

INTERVENTIONS:
Drug: Immune checkpoint inhibitor (ICI) — Immune checkpoint inhibitors included were targeting either PD-1, PD-L1 or CTLA-4, and had received FDA approval at the time of study (ATC classification): Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32), and Cemiplimab (L01XC33).
  Other Names: Ipilimumab (Yervoy, L01XC11); Nivolumab (Opdivo, L01XC17); Pembrolizumab (Keytruda, L01XC18); Durvalumab (Imfinzi, L01XC28); Avelumab (Bavencio, L01XC31); Atezolizumab (Tecentriq, L01XC32); Cemiplimab (Libtayo, L01XC33)

SUMMARY:
Immune checkpoint inhibitors (ICIs) are associated with a wide variety of cutaneous immune-related adverse events (cirAEs). These cirAEs are reported to be the most common immune-related adverse events (irAEs) and the first to appear. This study examines the appearance of cirAEs within the World Health Organization (WHO) pharmacovigilance database, VigiBase.

DETAILED DESCRIPTION:
ICIs have revolutionized clinical oncologic care. The ICIs that are currently FDA approved fall into three main categories: those that block the cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4; ipilimumab), block the programmed cell death protein-1 (anti-PD-1; nivolumab, pembrolizumab, cemiplimab), and block the programmed cell death ligand-1 (anti-PD-L1; atezolizumab, avelumab, durvalumab) pathway. There is a considerable diversity of cirAEs that have been reported with these ICIs in both monotherapy and combination therapy.

VigiBase is the WHO pharmacovigilance database that monitors individual case safety reports associated with certain drugs. The largest database of its kind in the world, VigiBase is managed by the Uppsala Monitoring Center (UMC) in Sweden, and since its inception in 1967 has received over 19 million individual case safety reports (ICSRs) from over 130 contributing countries. In this study, the investigators examine the appearance of cutaneous immune related adverse events in the setting of immunotherapy within VigiBase.

ELIGIBILITY:
Inclusion Criteria:

* Treated with either Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32), and Cemiplimab (L01XC33).
* Developed an adverse reaction that was submitted to a pharmacovigilance center and was determined to be related to aforementioned immune checkpoint inhibitors.
* Adverse reaction was determined to be within the System Organ Class (SOC) "Skin and subcutaneous disorder".

Exclusion Criteria:

* Adverse event was determined not to be immune-related (for example, infectious etiology) or was a symptom (e.g., edema).
* Adverse event developed before the administration of ICI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with an immune checkpoint inhibitor for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2214 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Cutaneous toxicity of ICIs | From 01/01/2008 to 08/31/2020
  Number of reported adverse events associated with ICIs within the Systems Organ Class (SOC) "Skin and subcutaneous disorders" with one of the 7 FDA-approved ICIs Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32), or Cemiplimab (L01XC33), alone or in any combination with each other.

SECONDARY OUTCOMES:
Reporting odds ratio for monotherapy vs combination therapy | From 01/01/2008 to 08/31/2020
  Reporting odds ratio for appearance of cirAEs, comparing the odds of appearance of cirAEs with monotherapy with PD-1, PD-L1, or CTLA-4 against combination therapy with a PD-1/PD-L1 and CTLA-4 agent.
Reporting odds ratio for differing monotherapy | From 01/01/2008 to 08/31/2020
  Reporting odds ratio for appearance of cirAEs comparing monotherapy with PD1 or PD-L1 against monotherapy with CTLA-4
Co-occuring irAEs | From 01/01/2008 to 08/31/2020
  Prevalence (%) of co-occuring irAEs within other organ systems (GI, endocrine/metabolic, pulmonary, cardiac, renal, hematologic, neurologic, rheumatologic, and ophthalmologic) with cirAEs.
Disproportionality assessment of cirAEs with ICIs | From 01/01/2008 to 08/31/2020
  Information component (IC), a Bayesian confidence neural network propagation method devised by the Uppsala Monitoring Center, will determine significant disproportionate signal of cirAEs associated with ICIs if >0 at the bottom of the 95% confidence interval (IC025 > 0).
Indication | From 01/01/2008 to 08/31/2020
  Prevalence (%) of malignancy types (such as melanoma, pulmonary, and renal cell carcinoma) for patients receiving ICIs and developing cirAEs.
Time to onset | From 01/01/2008 to 08/31/2020
  Time to onset of cirAEs after ICI administration, measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Kwatra, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Care Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le TK, Brown I, Goldberg R, Taylor MT, Deng J, Parthasarathy V, Bordeaux ZA, Alphonse MP, Kwatra MM, Naranbhai V, Gusev A, Alhariri J, LeBoeuf NR, Reynolds KL, Cappelli LC, Naidoo J, Brahmer JR, Kang S, Semenov YR, Kwatra SG. Cutaneous Toxicities Associated with Immune Checkpoint Inhibitors: An Observational, Pharmacovigilance Study. J Invest Dermatol. 2022 Nov;142(11):2896-2908.e4. doi: 10.1016/j.jid.2022.04.020. Epub 2022 May 20. PMID 35605659